CLINICAL TRIAL: NCT02903927
Title: Prospective Comparative Randomized Clinical Trial to Evaluate the Visual Performance of Two Monofocal Intraocular Lenses
Brief Title: Clinical Trial to Evaluate the Visual Performance of Two Monofocal Intraocular Lenses
Acronym: LUCIOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CT LUCIA 601PY BER 401-14
Record Dates: First submitted 2016-09-09; First posted 2016-09-16 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Catartact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT LUCIA (Experimental)
  Interventions: Device: Implantation of CT LUCIA IOL
- Acrysof IQ Sn60WF (Active Comparator)
  Interventions: Device: Implantation of Acrysof IQ SN60WF IOL

INTERVENTIONS:
Device: Implantation of CT LUCIA IOL
  Arms: CT LUCIA
Device: Implantation of Acrysof IQ SN60WF IOL
  Arms: Acrysof IQ Sn60WF

SUMMARY:
The main objective of the clinical study is to evaluate the performance of the CT LUCIA 601 PY for the monocular uncorrected distance visual acuity and compare it to the reference monofocal IOL Acrysof IQ SN60WF.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent;
* Patients of any gender, aged 50 to 90 years;
* Senile cataract in at least 1 eye;
* Assured follow-up examinations;
* Healthy eyes besides clinically significant cataract
* Biometry measurement/cataract density compatible with the IOLMaster evaluation.

Post-operative inclusion criteria:

* IOL implanted in the capsular bag;
* The IOL model (CT LUCIA 601PY or Acrysof IQ SN60WF) has been implanted;
* No intraoperative complications; no damaged capsular bag, no intraocular hemorrhage; no can opener rhexis.

Exclusion Criteria:

* • Patients unable to meet the limitations of the protocol or likely of non-cooperation during the trial;

  * Patients whose freedom is impaired by administrative or legal order;
  * Current participation in another drug or device investigation;
  * Allergy to heparin
  * Monophthalmic patient
  * Ocular disorders, other than cataract, that could potentially cause future acuity loss to a level of 0.20 logMAR (best-corrected) or worse the operated eye
  * Any anterior segment pathology that could significantly affect outcomes (e.g. chronic uveitis, iritis, corneal dystrophy, etc.)
  * Diabetic retinopathy
  * Traumatic cataract
  * Aniridia
  * Microphthalmus
  * Amblyopia
  * Degenerative visual disorders (e.g. macular degeneration, optic nerve atrophy, or retinal disorders)
  * Patient expected to require retinal laser treatment before the end of the follow-up
  * Previous intraocular and corneal surgery
  * Expected postop. astigmatism greater than 1 D
  * Any type of corneal disorder
  * Dementia
  * Diabetes mellitus
  * Pseudoexfoliation syndrome (PXF)
  * Glaucoma or IOP higher than 24mmHg under ocular hypertension treatment
  * Any other pathology or condition presenting, according to the investigator opinion, a risk for the patient

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity (UCVA) (monocular) | 6 months